CLINICAL TRIAL: NCT03685279
Title: Testing the Efficacy of the Nurtured Heart Approach: A Randomized Controlled Trial
Brief Title: Efficacy of the Nurtured Heart Approach to Reduce ADHD Behaviors in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Velia Nuno, Assistant Professor, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1707672022
Record Dates: First submitted 2018-08-28; First posted 2018-09-26 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2018-09

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NHA Group (Experimental): Six-week, online intervention with weekly, sequential, content knowledge and skills practice. Each week included recorded, slide presentations (narrated by the developer of the NHA, Howard Glasser); readings from "The Transforming the Intense Child Workbook" by Howard Glasser with Melissa Lowenstein; participants' skills practice, web postings, and live sessions with Howard Glasser and Advanced NHA Trainers.
  Interventions: Behavioral: Nurtured Heart Approach
- Control Group (Other): The Control Group received the same intervention after the collection of NHA Group post-intervention surveys.
  Interventions: Behavioral: Nurtured Heart Approach

INTERVENTIONS:
Behavioral: Nurtured Heart Approach — Based on three stands designed to reduce negative reactivity from parents/guardians, increase positive interactions, and set firm, clear limits.

SUMMARY:
This study evaluates the efficacy of the Nurtured Heart Approach (NHA) to reduce inattention and hyperactivity and impulsivity in children ages 6 - 8 years. Participants are parents or guardians of children diagnosed with, or suspected of, attention deficit hyperactivity disorder (ADHD). Participants are randomized into the immediate (NHA) or delayed (Control) group.

DETAILED DESCRIPTION:
The American Academy of Pediatrics recommends evidence-based parent and/or teacher behavioral therapy and/or medication to treat ADHD. A systematic review by Coates and colleagues found behavioral interventions decreased ADHD behaviors in children. The NHA is an intervention designed to teach parents a set of skills and attitudes to decrease ADHD in children. It has been applied in a number of settings from homes, schools, and foster care agencies both in several states in the U.S. and in over 16 countries. While widely accepted, the Approach has not been evaluated using scientifically rigorous methods.

ELIGIBILITY:
Inclusion Criteria:

* Parent or guardian of a child diagnosed with ADHD or suspected of ADHD
* Child must be 6 - 8 years of age
* Access to a computer with Internet

Exclusion Criteria:

* Child with ADHD, or suspected of ADHD, cannot have a diagnosis of autism

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Inattention | Six-week change from pre-intervention inattention to post-intervention inattention.
  Parent reported measure called Conners-3 Parent Short Form. Raw scores are converted into standardized T-scores using age- and sex-specific conversion standards. The minimum T-score is 40 and the maximum is 90. The six content subscales are inattention, hyperactivity/impulsivity, learning problems, executive function, defiance/aggression, and peer relations. Higher T-scores are worse.
Hyperactivity/Impulsivity | Six-week change from pre-intervention hyperactivity/impulsivity to post-intervention hyperactivity/impulsivity.
  Parent reported measure called Conners-3 Parent Short Form. Raw scores are converted into standardized T-scores using age- and sex-specific conversion standards. The minimum T-score is 40 and the maximum is 90. The six content subscales are inattention, hyperactivity/impulsivity, learning problems, executive function, defiance/aggression, and peer relations. Higher T-scores are worse.

SECONDARY OUTCOMES:
Parental Stress | Six-week change from pre-intervention parental stress to post-intervention parental stress.
  Parent reported measure called Parenting Stress Index - 4 Short Form. Scores are summed. A minimum raw score possible is 36 and maximum is 180. Higher values are worse.
Parenting Competency | Six-week change from pre-intervention parenting competency to post-intervention parenting competency.
  Parent reported measure called Parenting Sense of Competence. Scores are summed. A minimum score possible is 16 and maximum is 96. Higher value is a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No